CLINICAL TRIAL: NCT01416948
Title: Randomized Controlled Trial of Galantamine, Methylphenidate, and Placebo for the Treatment of Cognitive Symptoms in Patients With Traumatic Brain Injury (TBI) and/or Posttraumatic Stress Disorder (PTSD)
Brief Title: Cognitive REmediation After Trauma Exposure Trial = CREATE Trial
Acronym: CREATE
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: The funding agency, DoD, determined that the study could not meet its enrollment numbers by the end of the grant.
Sponsor: INTRuST, Post-Traumatic Stress Disorder - Traumatic Brain Injury Clinical Consortium (Other)
Collaborators: U.S. Army Medical Research and Development Command (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: INTRuST-CREATE
Record Dates: First submitted 2011-08-12; First posted 2011-08-15 (Estimated); Last update posted 2013-04-26 (Estimated); Status verified 2013-04

CONDITIONS: Posttraumatic Stress Disorder; Traumatic Brain Injury
Keywords: Cognitive Complaints, TBI, PTSD
MeSH Terms: conditions — Stress Disorders, Post-Traumatic; Brain Injuries, Traumatic | interventions — Methylphenidate; Galantamine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Sugar Pill (Placebo Comparator)
  Interventions: Drug: Placebo Capsule
- Galantamine (Active Comparator)
  Interventions: Drug: Galantamine 12 mg
- Methylphenidate (Experimental)
  Interventions: Drug: Methylphenidate Hydrochloride 20 mg

INTERVENTIONS:
Drug: Methylphenidate Hydrochloride 20 mg — For patients assigned to the MPH arm of the study, the drug will be initiated at 5 mg bid at week 0, and increased to 10 mg bid at week 4, and finally increased to 20 mg bid at week 8 and then held constant until the major outcome assessment at week 12. The drug will be gradually tapered during weeks 12-14. If adverse events ensue, the subject's dose can be held at the current dose (rather than proceeding with scheduled dose increases) or reduced to the previous dose. Subjects who cannot tolerate the minimum dose (5 mg bid) will be withdrawn from the study.
  Other Names: Ritalin
  Arms: Methylphenidate
Drug: Placebo Capsule — For patients randomly assigned to the placebo arm of the study, placebo will be administered BID at Week 0 through Week 12. Matching placebo will be administered to match the taper period.
  Arms: Sugar Pill
Drug: Galantamine 12 mg — For patients randomly assigned to the GAL arm of the study, the drug will be initiated at 4 mg bid at week 0, increased to 8 mg bid at week 4, and finally increased to 12 mg bid at week 8 and then held constant until the major outcome assessment at week 12. The drug will be gradually tapered during weeks 12-14. If adverse events ensue, the subject's dose can be held at the current dose (rather than proceeding with scheduled dose increases) or reduced to the previous dose. Subjects who cannot tolerate the minimum dose (4 mg bid) will be withdrawn from the study.
  Other Names: Razadyne
  Arms: Galantamine

SUMMARY:
This study will evaluate the efficacy of methylphenidate and galantamine in the treatment of persistent cognitive symptoms associated with posttraumatic stress disorder (PTSD) and/or traumatic brain injury (TBI).

DETAILED DESCRIPTION:
Both traumatic brain injury (TBI) and posttraumatic stress disorder (PTSD) are prevalent in service members returning from Operation Enduring Freedom, Operation Iraqi Freedom, and Operation New Dawn (OEF/OIF/OND). Virtually all individuals who suffer TBI (TBI) have acute cognitive effects, and a significant number have persistent symptoms. A large number of individuals with PTSD also report problems with cognition, however, little is known about the treatment of cognitive complaints in either condition and less is known about cognitive complaints in individuals with co-occurring TBI and PTSD.

There is some preclinical evidence that both the cholinergic and catecholaminergic neurotransmitter systems play important roles in cognitive function in healthy individuals as well as those with mTBI and/or PTSD. We propose to evaluate the efficacy of two pharmacotherapies, one that predominantly augments cholinergic function (galantamine [GAL]) and one that augments predominantly catecholaminergic function (methylphenidate [MPH]), for reducing cognitive symptoms in individuals with TBI and/or PTSD.

Using a double-blind, randomized, placebo controlled design, 159 individuals with TBI and/or PTSD with persistent cognitive complaints will be randomized to receive galantamine 12 mg BID, methylphenidate 20 mg BID, or placebo for 12 weeks. The primary objective is to assess the efficacy of galantamine and methylphenidate in reducing cognitive complaints in patients with PTSD and/or TBI. Secondary objectives are to assess the extent to which non-cognitive distress responds to galantamine or methylphenidate, and assess the effect that galantamine and methylphenidate have on cognitive performance.

ELIGIBILITY:
Inclusion Criteria:

1. Aged 18-55 years
2. Has a DSM-IV diagnosis of chronic (≥ 3 months duration) PTSD and/or a history of TBI (≥ 3 months duration) as established by the INTRuST standard TBI Screening questionnaire.
3. TBI must have occurred ≥ 90 days prior to the screening visit
4. With either diagnosis (i.e., PTSD or TBI), the subject must have clinically significant cognitive complaints, as indicated by a T score ≥ 60 on the postmorbid Cognitive scale of the RNBI
5. Interested in receiving treatment for cognitive symptoms
6. Capable of giving informed consent

Exclusion Criteria:

1. Known sensitivity, or previous adverse reaction(s), to GAL or other acetylcholinesterase inhibitors such as donepezil or rivastigmine OR Known sensitivity or previous adverse reactions to MPH or other stimulant medications (e.g., dextroamphetamine, long-acting methylphenidate preparations)
2. Pregnant, likely to become pregnant, or lactating (female subjects only)
3. Does not speak English
4. WRAT scaled score < 70
5. History of glaucoma
6. History of cardiac conditions (e.g., bradycardia, AV block) or history of taking medications that are associated with conduction abnormalities
7. History of seizure disorder (including post-traumatic epilepsy), neurosurgery, or neurodisability [Note that history of "impact seizure" is permitted]
8. Lifetime history of psychotic disorder, Bipolar I, stimulant abuse or dependence, or tic disorder
9. Alcohol dependence, alcohol abuse*, substance abuse, or substance dependence in the past 6 months [*Alcohol abuse will be defined as MINI diagnosis of "Alcohol Abuse" AND an AUDIT-C score of ≥ 5; Dawson, Grant, & Stinson, 2005].
10. Current active suicidal ideation, or history of actual attempt within the past 10 years
11. Current severe depressive symptoms, as indicated by a score of 20 or higher on the PHQ-9
12. Current (or past 2-week) use of monoamine oxidase inhibitors [Washout period of at least 2 weeks is required]
13. Current (or past 2-week) use of medications that potentiate cholinergic function (i.e., other cholinesterase inhibitors or procholinergic agents), or use of over-the-counter procholinergics [Washout period of at least 2 weeks is required]
14. Current (or past 2-week) use of amphetamine-type stimulants or modafinil
15. Current use of any other psychotropic medication that fails to meet the stabilization criterion of a minimum of 4 weeks on the same medication(s) and dose(s)
16. Prior use of any other psychotropic medication that fails to meet the washout criterion of 2 weeks
17. Concurrent cognitive therapy, that will not be discontinued at least 7 days prior to the baseline visit
18. Baseline ECG and/or bloodwork reveals serious illness that precludes participation or use of study medications
19. Any procedure requiring general anesthesia
20. History of peptic ulcer disease or GI bleed or endoscopic procedure for GERD within the last year. Subjects taking physician prescribed treatment for GERD will be allowed to participate at the discretion of the PI after discussion with the primary treating physician.
21. Current (or past 2-week) use of alpha 2 adrenergic agonists such as guanfacine

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 32 (Actual)
Dates: Start 2011-08; Primary Completion 2013-03 (Actual); Study Completion 2013-03 (Actual)

PRIMARY OUTCOMES:
Ruff Neurobehavioral Inventory - Postmorbid Cognitive Scale | Baseline through Week 12
  The Ruff Neurobehavioral Inventory (RNBI; Ruff & Hibbard, 2003) is a self-report instrument for assessment of a wide range of symptoms (cognitive, emotional, and physical), as well as quality of life and daily functioning. It was designed to assess these areas in individuals who have recently been affected by an injury, illness, or other stressor. The Postmorbid Cognitive scale will be used as the primary outcome measure in this study. The Postmorbid Cognitive scale consists of 24 items assessing Attention/Concentration, Executive Functions, Learning/Memory, and Speech/Language.

SECONDARY OUTCOMES:
Rivermead Postconcussion Symptom Questionnaire (RPCSQ) | Baseline through week 12
  The RPCSQ (N King, 1995), which can be self-administered or given by an interviewer, asks patients to rate the severity of 16 different symptoms commonly found after a mild traumatic brain injury. Patients are asked to rate the severity of each symptom over the past week and compare to the severity before their injury. This instrument will be used to determine the extent to which the broad spectrum of TBI symptoms respond to GAL and MPH.
Patient Health Questionnaire-9 (PHQ - 9) | Baseline through week 12
  The PHQ - 9 (Pfizer, 1999) is the self-administered 9 item depression scale of the Patient Health Questionnaire. This instrument will be used to determine the extent to which GAL and MPH improve depressive symptoms in participants with PTSD and/or TBI.
PTSD Checklist - Specific Event Version (PCL-S) | Baseline through week 12
  The PTSD Checklist - Specific Event Version (Weathers, 1993) is a 17 item self-report measure of DSM IV symptoms of PTSD in response to a specific event, used for screening and diagnosis of PTSD and monitoring symptom change during treament. This measure will be used to determine the extent to which the broad spectrum of PTSD symptoms responds to GAL and MPH.
PreMorbid-Postmorbid Difference Score on Cognitive Scale of Ruff Neurobehavioral Inventory | Baseline through 12 weeks
  This measurement will be used to determine the extent to which GAL and MPH reduce the perceived difference between subjects' premorbid and postmorbid cognitive functioning.
Neuropsychological Tests of Memory, Attention and Other Executive Functions | Baseline through 12 weeks
  These measurements will be used to determine the extent to which GAL and MPH affect objective cognitive functioning in participants with PTSD and/or TBI as measured on the following neuropsychological tests: Rey Verbal Auditory Learning Test; Trail Making Test; WAIS-III Processing Speed Index and Digit Span; Digit Vigilance test; WMS-III Letter-Number Sequencing; Brief Visuospatial Memory Test-Revised; Paced Auditory Serial Addition Test; Continuous Performance Test; and D-KEFS Verbal Fluency.

CONTACTS AND LOCATIONS:
Overall Officials: Thomas W McAllister, M.D., Principal Investigator — Dartmouth-Hitchcock Medical Center; Ross Zafonte, M.D., Principal Investigator — Spaulding Rehabilitation Hospital
Locations (7):
- United States (7):
  - VA San Diego Healthcare System, San Diego, California
  - Spaulding Rehabilitation Hospital, Boston, Massachusetts
  - Manchester VA Medical Center, Manchester, New Hampshire
  - Duke University, Durham, North Carolina
  - University of Cincinnati, Cincinnati, Ohio
  - Ralph H. Johnson VA Medical Center, Charleston, South Carolina
  - White River Junction VA Medical Center, White River Junction, Vermont